CLINICAL TRIAL: NCT05334251
Title: General Anesthesia or Combined Spinal-epidural Anesthesia With Ketofol Sedation in Colon Cancer Surgery?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ayça Özcan, Associate Professor, MD, Ankara City Hospital Bilkent
Other Study IDs: E2-21-1021
Record Dates: First submitted 2021-11-19; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Colon Cancer; Anesthesia
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- general anesthesia group: Patients in this group will undergo open colon cancer surgery under general anesthesia. Epidural catheterization will be applied for postoperative analgesia.
- combined spinal-epidural anesthesia group: Patients in this group will undergo open colon cancer surgery under combined spinal-epidural anesthesia with ketofol sedation. Epidural catheterization will be applied for postoperative analgesia.
  Interventions: Other: combined spinal-epidural anesthesia

INTERVENTIONS:
Other: combined spinal-epidural anesthesia — Combined spinal and epidural anaesthesia is a regional anaesthetic technique, which combines the benefits of both spinal anaesthesia and epidural anaesthesia and analgesia. The spinal component gives a rapid onset of a predictable block. The indwelling epidural catheter gives the ability to provide long lasting analgesia and to titrate the dose given to the desired effect.
  Groups: combined spinal-epidural anesthesia group

SUMMARY:
Anesthesia management in colon cancer surgery affects the postoperative mobilization, discharge and oral intake times of the patients. Due to the side effects of opioids, their use is tried to be reduced and therefore regional anesthesia methods are preferred in suitable patients. Especially in the preoperative period, opioid use has a negative effect on the recovery processes, morbidity and mortality of the patients. Epidural analgesia, a central block method, is recommended for postoperative pain control in ERAS protocols. Opioids suppress cellular and humoral immunity. Epidural analgesia reduces both opioid consumption and surgical stress response. It has been shown that epidural analgesia maintains the immune functions of patients and is associated with a decrease in tumor recurrence. It has also been shown to reduce postoperative pain, hypercoagulability and pulmonary complications, increase exercise capacity and accelerate the return of intestinal functions to normal. In line with this information, in this study, it was aimed to investigate the differences in the postoperative period in patients managed with regional anesthesia.

In the study, it was planned to create two groups who underwent open surgery for colon cancer. The first group will be operated under general anesthesia and the second group will be operated under combined spinal-epidural anesthesia with ketofol sedation. An epidural catheter will be inserted in both groups for postoperative pain management. In the study, patients' age, gender, weight, comorbidity, ASA score, amount of local anesthetic used, postoperative VAS scores, mobilization time, time to start oral intake, nasogastric withdrawal time, drain removal time, urinary catheter withdrawal time, hospitalization time and total cost will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 40 years of age who are scheduled for open surgery with a diagnosis of colon cancer

Exclusion Criteria:

* Local anesthetic allergy
* Patients scheduled for laparoscopic surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 40 years of age who are scheduled for open surgery with a diagnosis of colon cancer.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) | postoperative 2nd hour.
  A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 5 cm horizontal line (between 0 and 5 points, 0 meaning 'no pain' and 5 meaning the worst) and this rating is then measured from the left edge (=Visual Analog Scale score).
visual analog scale (VAS) | postoperative 4th hour.
  A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 5 cm horizontal line (between 0 and 5 points, 0 meaning 'no pain' and 5 meaning the worst) and this rating is then measured from the left edge (=Visual Analog Scale score).
visual analog scale (VAS) | postoperative 8th hour.
  A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 5 cm horizontal line (between 0 and 5 points, 0 meaning 'no pain' and 5 meaning the worst) and this rating is then measured from the left edge (=Visual Analog Scale score).
visual analog scale (VAS) | postoperative 12th hour.
  A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 5 cm horizontal line (between 0 and 5 points, 0 meaning 'no pain' and 5 meaning the worst) and this rating is then measured from the left edge (=Visual Analog Scale score).
visual analog scale (VAS) | postoperative16th hour.
  A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 5 cm horizontal line (between 0 and 5 points, 0 meaning 'no pain' and 5 meaning the worst) and this rating is then measured from the left edge (=Visual Analog Scale score).
visual analog scale (VAS) | postoperative 24th hour.
  A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 5 cm horizontal line (between 0 and 5 points, 0 meaning 'no pain' and 5 meaning the worst) and this rating is then measured from the left edge (=Visual Analog Scale score).
time to start oral intake | to be observed until the start of oral intake after the operation. it will be assessed up to 720 hours.
  the time the patient start to consume orally after the operation
mobilization time | to be observed until the start of walking after the operation. it will be assessed up to 720 hours.
  the time the patient was start to walk after the operation
urinary catheter withdrawal time | to be observed until the withdrawal of urinary catheter after the operation. it will be assessed up to 720 hours.
  the time the urinary catheter was withdrawn after the operation
hospitalization time | from hospitalization for the operation to the day of discharge, it will be assessed up to 30 days.
  The time from the day the patient was hospitalized before the operation to the day of discharge after the operation.
nasogastric withdrawal time | to be observed until the withdrawal of nasogastric tube after the operation. it will be assessed up to 720 hours.
  the time the nasogastric tube was withdrawn after the operation.
drain removal time | to be observed until the withdrawal of abdominal drain after the operation. it will be assessed up to 720 hours.
  the time the abdominal drain was withdrawn after the operation.
complications | to be observed for 30 days postoperatively.
  all complications related with surgery or anesthesia
blood pressure | preoperatively
  patients' mean arterial pressure levels
blood pressure | perioperatively. "30 minutes" will be taken as the measurement period.
  patients' mean arterial pressure levels
FiCO2 | preoperatively
  inspiratory carbondioxide level
FiCO2 | perioperatively. "30 minutes" will be taken as the measurement period.
  inspiratory carbondioxide level
sPO2 | preoperatively
  oxygene saturation
sPO2 | perioperatively. "30 minutes" will be taken as the measurement period.
  oxygene saturation

REFERENCES:
- [Background] Wu HL, Tai YH, Mandell MS, Tsou MY, Yang SH, Chen TH, Chang KY. Effect of epidural analgesia on cancer prognosis after colon cancer resection: a single-centre cohort study in Taiwan. BMJ Open. 2020 Oct 22;10(10):e036577. doi: 10.1136/bmjopen-2019-036577. PMID 33093029
- [Background] Cummings KC III, Zimmerman NM, Maheshwari K, Cooper GS, Cummings LC. Epidural compared with non-epidural analgesia and cardiopulmonary complications after colectomy: A retrospective cohort study of 20,880 patients using a national quality database. J Clin Anesth. 2018 Jun;47:12-18. doi: 10.1016/j.jclinane.2018.03.005. Epub 2018 Mar 12. PMID 29544203
- [Background] Ljungqvist O, Hubner M. Enhanced recovery after surgery-ERAS-principles, practice and feasibility in the elderly. Aging Clin Exp Res. 2018 Mar;30(3):249-252. doi: 10.1007/s40520-018-0905-1. Epub 2018 Feb 16. PMID 29453605
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190

DOCUMENTS (1):
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT05334251/ICF_000.pdf